CLINICAL TRIAL: NCT06760598
Title: Evaluation of the Relationship Between Thoracic Kyphosis and Quadriceps Muscle Thickness with Balance and Fall Risk in Women with Postmenopausal Osteoporosis
Brief Title: Evaluation of Balance and Functionality in Postmenopausal Osteoporosis Using Quadriceps Femoris Muscle Thickness, Beyond Thoracic Hyperkyphosis
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eslem Peker Belene, Medical Doctor, Istanbul University - Cerrahpasa
Other Study IDs: E-83045809-604.01.01-439462
Record Dates: First submitted 2024-12-27; First posted 2025-01-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis; Sarcopenia; Ultrasonography; Hyperkyphosis
Keywords: muscle thickness; sarcopenia; hyperkyphosis; ultrasonography
MeSH Terms: conditions — Osteoporosis; Sarcopenia; Kyphosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To determine the impact of thoracic hyperkyphosis, sarcopenia and quadriceps muscle thickness evaluated by ultrasonography (USG) on balance, fall risk and functional parameters in women with postmenopausal osteoporosis, to assess their interrelationships and to compare the clinical characteristics of sarcopenia and thoracic hyperkyphosis.

DETAILED DESCRIPTION:
An observational study was conducted on patients with PMO and/or osteoporotic vertebral fractures according to WHO criteria. One hundred seventeen patients who were 50 years of age or older, with a diagnosis of PMO and/or osteoporotic vertebral fractures according to WHO criteria, who were able to ambulate without any assistive devices were included in the study. Patients with a history of neurological disease which may affect balance and proprioception, visual and vestibular disease, previous major lower extremity surgery or previous vertebra surgery were excluded. The investigators also excluded the patients with advanced heart, liver, or renal failure, stage 4 knee osteoarthritis, psychiatric disorders, and use of any medication affecting the central nervous system.

Age, height, weight, body mass index (BMI), comorbidities, medications, previous surgeries, steroid use, previous fractures and the energy level of these fractures (low or high), fracture location, family history of fractures, alcohol use, smoking, menopausal age and the number of falls in a year were questioned. The FRAX algorithm was used to determine the risk of fracture.

The Cobb angle of thoracic kyphosis was calculated radiographically and QFM thickness was measured from anterior thigh via ultrasonography (USG). The presence of sarcopenia was determined. Balance, fall risk and physical function were evaluated with tandem stance and gait test, Berg balance scale (BBS), Timed up and go test (TUG), hand grip strength, chair stand test (CST).

ELIGIBILITY:
Inclusion Criteria:

* Patient who were 50 years of age or older, had postmenopausal osteoporosis and/or osteoporotic vertebral fractures according to WHO criteria,
* Patient who were able to ambulate without any assistive devices

Exclusion Criteria:

* History of neurological disease which may affect balance and proprioception,
* Visual and vestibular disease
* Previous major lower extremity surgery or previous vertebra surgery
* Advanced heart, liver, or renal failure
* Stage 4 knee osteoarthritis
* Psychiatric disorders
* Use of any medication affecting the central nervous system.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with Postmenopausal Osteoporosis
Study Population: Patients aged 50 years and over with postmenopausal osteoporosis and/or osteoporotic vertebral fractures according to WHO criteria who applied to the outpatient clinic of the Department of Physical Medicine and Rehabilitation, Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
tandem stance and gait test | Data were collected over a single measurement period of 6 months.
  static and dynamic balance was measured.
berg balance scale | Data were collected over a single measurement period of 6 months.
  Berg balance scale was originally developed for the assessment of postural control and is widely used in many areas of rehabilitation. There are 14 items in the scale, like commonly performing in daily activities sitting and standing balance, transfers, turning, and retrieving objects from the floor. The highest total score is 56 points. If the patient scores between 0-20 points, they are considered wheelchair dependent, between 21-40 points they can walk with assistance and between 41-56 points they are considered independent in mobilization activities.
Timed up and go test | Data were collected over a single measurement period of 6 months.
  There is a significant relationship between TUG times and functional mobility level
chair stand test | Data were collected over a single measurement period of 6 months.
  The five times CST evaluates the strength, power, and endurance of the lower extremity muscle group, particularly the quadriceps femoris muscle
quadriceps femoris muscle thickness | Data were collected over a single measurement period of 6 months.
  evaluated by ultrasound
thoracic kyphosis | Data were collected over a single measurement period of 6 months.
  The lateral thoracic vertebra radiographs were taken while standing position, the Cobb angle was automatically obtained by computer-aided method by marking the parallel lines drawn from the upper edge of the upper thoracic vertebra (T4), and the lower edge of the lower thoracic vertebra (T12)

CONTACTS AND LOCATIONS:
Overall Officials: ESLEM PEKER BELENE, Principal Investigator — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty; ZEYNEP ÜLKÜ AKARIRMAK, Study Director — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty; RANA TERLEMEZ, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty; OSMAN AYKAN KARGIN, Study Chair — Istanbul University- Cerrahpasa, Cerrahpasa Medical Faculty
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University Cerrahpasa, Istanbul, Istanbul
  - Istanbul University Cerrahpasa, Cerrahpasa Medical Faculty, Istanbul, SÜLEYMANPAŞA

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months after publication of primary results
Access Criteria: Academic and Clinical Researchers, Regulatory Authorities and Non-commercial Researchers and Public Health Organizations can access the data Demographic and Clinical Data, Outcome Measures,Study protocols, statistical analysis plans, and publications can be accessed Submit a Request, Approval Process, Secure Access will be accessed